CLINICAL TRIAL: NCT06427408
Title: Cellular Transcriptomic Trajectory of the Human Placenta During Pregnancy
Brief Title: Longitudinal Study of Gene Expression in the Human Placenta During First-trimester and Full-term Pregnancy at the Single Cell Level
Acronym: VilliRNAseq
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240045; 2022-A02452-41 (Other: France : Ministry of Health)
Record Dates: First submitted 2024-05-16; First posted 2024-05-23 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Related
Keywords: Placenta; Single nuclei RNA-seq; Preeclampsia; Pregnancy outcomes
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Placental tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Villi RNASeq: There is only one study group : patients with placental transcriptomic analysis by single nucleus RNA-seq approach
  Interventions: Other: Non applicable

INTERVENTIONS:
Other: Non applicable — Placental transcriptomic analysis

SUMMARY:
The single nucleus RNA-seq approach allows the placental transcriptome to be analyzed from nuclei, thus preserving the integrity of placental syncytium. This approach is feasible on small fragments of villi and offers for the first time the possibility to consider the characterization of gene expression within the structural unit of the human placenta during pregnancy (at the 1st trimester and childbirth)

DETAILED DESCRIPTION:
Chorionic villus biopsies are routinely performed between 11SA and 15SA at the Fetal Medicine Unit́ of the Port-Royal Maternity Hospital (CPDPN Cochin) after the patient has signed an information and consent form for the genetic analysis.

The patient will be asked to participate to the VilliRNAseq project and will sign the consent form of the study. After the cytogeneticist observation, a villi fragment will be snap-frozen in liquid nitrogen and stored at -80°C until use. Each patient sampled in the first trimester is followed until the end of the pregnancy. At delivery, cesarean section or vaginal delivery, a placental sample will be snap-frozen in liquid nitrogen and stored at -80°C until use.

Isolation, sorting and encapsidation of nuclei, RNA libraries preparation and sequencing will be carried out using 10x Genomics technology. State-of-the-art computational analyses to decipher trajectories and cell-to-cell communications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50
* Progressive monofoetal pregnancy between 11 and 15 weeks of amenorrhea
* Patient with prenatal medical indication and requesting chorionic villus biopsy with cytogenetic analysis or molecular genetics
* Patient scheduled for delivery at Port-Royal Maternity Hospital

Exclusion Criteria:

* Minor patient
* Multiple pregnancy
* Patient's objection
* Without health insurance
* Patient under guardianship or curatorship

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnancy
Study Population: Women in their pregnancy follow-up at the Maternité Port-Royal-Cochin
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Analysis of the cellular transcriptomic trajectory of the human placenta | Day 0
  Sequencing data will be analysed at the Institut Cochin, cell trajectories will be modelled and intracellular communications will be inferred
Analysis of the cellular transcriptomic trajectory of the human placenta | At childbirth
  Sequencing data will be analysed at the Institut Cochin, cell trajectories will be modelled and intracellular communications will be inferred

SECONDARY OUTCOMES:
Collection of placental samples | Day 0
Collection of placental samples | At childbirth
Identification of early markers of pregnancy complications | Until at Childbirth
  Pre-eclampsia, growth retardation in utero, delivery before 37 SA

CONTACTS AND LOCATIONS:
Overall Officials: Céline MÉHATS, PHD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Hélène COLLINOT, MD, Principal Investigator — APHP
Locations (1):
- Maternité Port-Royal, Cochin hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided